CLINICAL TRIAL: NCT02379091
Title: A 24-Week Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose Finding Study to Evaluate the Efficacy and Safety of 3 Doses of Namilumab (20 mg, 80 mg and 150 mg) in Combination With Methotrexate (MTX) in Subjects With Moderate to Severe Rheumatoid Arthritis (RA)
Brief Title: Dose Finding Study of Namilumab in Combination With Methotrexate in Participants With Moderate to Severe Rheumatoid Arthritis (RA)
Acronym: NEXUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M1-1188_202; U1111-1151-6931 (Registry Identifier: WHO); 2013-002805-76 (EudraCT Number); 14/SC/1252 (Registry Identifier: NRES); 153300410A0071 (Registry Identifier: RNEC); JapicCTI-152979 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-11-28; First posted 2015-03-04 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Drug therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — namilumab; Methotrexate; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Namilumab placebo-matching, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks for 12 weeks. Participants were assessed for response (a 20% improvement from Baseline in both swollen and tender joint counts). If the participant was a responder, the current treatment continued every 4 weeks up to Week 24. If the participant was a non-responder, the participant entered an open-label period and received namilumab 150 mg/mL, SC injection, every 4 Weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
  Interventions: Drug: Placebo; Drug: Methotrexate; Drug: Folic/folinic acid
- Namilumab 20 mg/mL (Experimental): Namilumab 20 mg/mL, subcutaneous (SC) injection, once on Days 1, 15, 43, 71 and every 4 weeks for 12 Weeks. Participants were assessed for response (a 20% improvement from Baseline in both swollen and tender joint counts). If the participant was a responder, the current treatment continued every 4 weeks up to Week 24. If the participant was a non-responder, the participant entered an open-label period and received namilumab 150 mg/mL, SC injection, every 4 Weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
  Interventions: Drug: Namilumab; Drug: Methotrexate; Drug: Folic/folinic acid
- Namilumab 80 mg/mL (Experimental): Namilumab 80 mg/mL, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks for 12 Weeks. Participants were assessed for response (a 20% improvement from Baseline in both swollen and tender joint counts). If the participant was a responder, the current treatment continued every 4 weeks up to Week 24. If the participant was a non-responder, the participant entered an open-label period and received namilumab 150 mg/mL, SC injection, every 4 Weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
  Interventions: Drug: Namilumab; Drug: Methotrexate; Drug: Folic/folinic acid
- Namilumab 150 mg/mL (Experimental): Namilumab 150 mg/mL, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks for 12 Weeks. Participants were assessed for response (a 20% improvement from Baseline in both swollen and tender joint counts). If the participant was a responder, the current treatment continued every 4 weeks up to Week 24. If the participant was a non-responder, the participant was discontinued from the study. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
  Interventions: Drug: Namilumab; Drug: Methotrexate; Drug: Folic/folinic acid

INTERVENTIONS:
Drug: Namilumab — Namilumab subcutaneous injection
  Arms: Namilumab 150 mg/mL; Namilumab 20 mg/mL; Namilumab 80 mg/mL
Drug: Placebo — Namilumab placebo-matching subcutaneous injection
  Arms: Placebo
Drug: Methotrexate — Methotrexate tablets
Drug: Folic/folinic acid — Folic/folinic acid tablets

SUMMARY:
The purpose of this study is to establish proof of concept and identify the optimal efficacious dose for namilumab in RA in patients with an inadequate response to methotrexate (MTX-IR) and in patients with an inadequate response to one tumor necrosis factor (TNF)-inhibitor (TNF-IR).

DETAILED DESCRIPTION:
The drug being tested in this study is called namilumab. Namilumab is being tested to treat rheumatoid arthritis (RA) in people who have an inadequate response to methotrexate, and in people who have an inadequate response to tumor necrosis factor-inhibitor (TNF-IR). This study will look at improvement in disease activity in participants who take namilumab.

The study will enroll approximately 100 patients. Participants will be randomly assigned (by chance) to one of the four treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Namilumab 20 mg/mL subcutaneous injection
* Namilumab 80 mg/mL subcutaneous injection
* Namilumab 150 mg/mL subcutaneous injection
* Placebo (dummy inactive subcutaneous injection) - this is a medication that looks like the study drug but has no active ingredient.

All participants will receive namilumab or placebo as specified in the protocol. A stable dose of methotrexate and daily folic acid will also be required treatments.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is up to approximately 40 weeks. Participants will make multiple visits to the clinic, including a follow-up assessment up to 18 weeks after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is male or female and aged 18 years (20 years in Japan) or older (65 years maximum in Czech Republic) at time of signing the informed consent form.
4. Must have adult onset rheumatoid arthritis (RA) as defined by the 2010 American College of Rheumatology (ACR)/ European League against Rheumatism (EULAR) criteria for the classification of RA for at least 6 months prior to Screening Visit.
5. Must have active disease defined as:

   a. At least moderately active disease defined by Disease Activity Score 28 based on C-reactive protein [DAS28(CRP)] ≥3.2 at screening and Disease Activity Score 28 based on Erythrocyte Sedimentation Rate [DAS28(ESR)] ≥3.2 at baseline visit [Day 1] and Swollen joint count (SJC) ≥4 (within the 28 joints from DAS28) at both the Screening and baseline [Day 1] Visits.
6. Visual analog scale (VAS) pain >40 mm as measured using the 100 mm study site electronic VAS scale at the Screening Visit and baseline [Day 1] Visits.
7. Currently receiving treatment for Rheumatoid Arthritis (RA) with methotrexate (MTX), and:

   * Has received MTX on a weekly basis for at least 3 months prior to the Baseline (Day 1) Visit AND;
   * Has received treatment with 15 mg/week ≤MTX ≤25 mg/week (6 mg/week ≤MTX ≤16 mg/week in Japan) at a stable dose via the same route of administration and formulation for at least 8 weeks prior to Baseline [Day 1] Visit

   OR:

   For participants outside Japan, a stable dose for at least 8 weeks of MTX of ≥7.5 mg/week is acceptable, if the MTX dose has been reduced for reasons of documented intolerance to MTX, e.g. hepatic or hematological toxicity documented in Electronic case report form (eCRF), or per local requirement.
8. Willing to continue or initiate treatment with oral folic acid (at least 5 mg/week) or equivalent and be treated during the entire study (mandatory co-medication for MTX treatment).
9. Must have a posterior, anterior (PA) and lateral chest x-ray obtained within 3 months prior to Screening, or recorded during screening.
10. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study until the end of the safety follow up (18 weeks after last dose).
11. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of the informed consent throughout the duration of the study until the end of the safety follow up (18 weeks after last dose).
12. Is able and willing to complete questionnaires at home using an electronic device in an approved language.
13. Has either Inadequate response to methotrexate (MTX-IR) or Inadequate response to TNF-inhibitor (TNF-IR).

Exclusion Criteria:

1. Participants <18 years of age (<20 years in Japan) or less than the legal adult age in the country of the study site, whichever is higher. Participants >65 years of age in Czech Republic.
2. Has received any investigational compound within 30 days, or within 5 half lives (whichever is longer) prior to the Screening Visit, or is participating or plans to participate in any other clinical study during this study.
3. Has a history of or currently has any inflammatory joint disease other than RA (eg, gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy or Lyme disease) or other systemic autoimmune disorder (eg, systemic lupus erythematosus [SLE], inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease or other overlap syndrome).
4. Has any major systemic features of RA, eg, Felty's syndrome, vasculitis or interstitial fibrosis of the lungs.
5. Has a diagnosis of primary fibromyalgia that would make it difficult to appropriately assess RA activity for the purposes of this study.
6. History of juvenile idiopathic arthritis or arthritis onset prior to age 16.
7. Is required to take or has taken excluded medications.

Has any of the following laboratory abnormalities at the screening visit (identified by the central laboratory):

1. Hemoglobin <8.5 g/dL;
2. Neutrophils <1500/mm^3;
3. Platelet count <75000 cells/mm^3;
4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN);
5. Bilirubin (total) >ULN, unless Gilbert's disease has been determined by genetic testing and has been documented.

   9. Has a history of hypersensitivity or allergies to any of the contents of the formulation.

   10. Has any clinically significant illness, including infection requiring antibiotics, within 4 weeks prior to the first dose of study medication, which may influence the outcome of the study.

   11. Has an underlying condition that predisposes to infections (eg, immunodeficiency, poorly controlled diabetes history, splenectomy).

   12. Evidence of clinically significant respiratory disease, on the basis of review the data from participants' respiratory assessments, including chest x-ray, lung function tests (forced expiratory volume in one second [FEV1] and forced vital capacity [FVC]) by spirometry performed at screening). The participants must have Saturation of peripheral oxygen (SpO2) ≥94%, FEV1 and FVC ≥60 % of predicted values and a Medical Research Council (MRC) Breathlessness Scale score of less than 4 at Screening and at Baseline and no uncontrolled lung disease. A participant's treatment which has been modified to control lung disease within 24 weeks prior to screening is exclusionary.

   13. History of clinically significant interstitial lung disease (ILD) eg, history of chronic or recurrent pulmonary infection where macrophages are important for the clearance of the infection eg, pneumocystis jiroveci pneumonia (PJP) formerly known as pneumocystis carinii pneumonia (PCP), allergic bronchopulmonary aspergillosis (ABPA), nocardia infections, Actinomyces infection, Japanese and Korean participants will be tested using Beta glucans test and participants will be excluded unless the Beta-Glucans test is negative.

   14. Presence or history of active tuberculosis (TB) or latent TB infection, where no anti-TB treatment has been given or where successful completion of an appropriate course of anti-TB therapy cannot be documented.

   15. A positive QuantiFERON-TB Gold test and/or evidence of active or latent TB by chest X-ray, not accompanied by initiation of an approved regimen of anti-TB therapy at least 12 months prior to the Baseline visit.

   16. Has a known history of infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus, or has serological findings at the Screening Visit which indicate active or latent hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.

   (Japan only) Participant has a positive result for hepatitis B virus surface antigen (HBsAg), hepatitis B virus antibody [hepatitis B surface antibody (HBs antibody) / hepatitis B virus core antibody (HBc antibody)], hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody. However, participants who are HBs antibody solely positive (but HBsAg and HBc antibody negative), resulting from hepatitis B virus (HBV) vaccination, are not to be excluded from the study.

   17. Has a history of severe chronic obstructive pulmonary disease (COPD) and/or history of severe COPD exacerbation(s), or a history of asthma with exacerbations requiring hospitalization (including emergency or acute care treatments), within the last 12 months prior to the Screening visit.

   18. History of MTX-associated lung toxicity. 19. Has a history or evidence of a clinically significant disorder (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric), condition or disease that, in the opinion of the investigator and/or Medical Monitor would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

   20. Any significant cardiac disease (eg, coronary artery disease with unstable angina, coronary heart failure New York Heart Association [NYHA] Class III and IV, familial long QT syndrome).

   21. Has a history of treatment with anti-chemotherapy (eg, alkylating agents, anti-metabolites [except MTX and Azathioprine], and purine analogues) and/or anti-cancer monoclonal antibodies within the last 5 years with the exception of topical anticancer drugs used in the treatment of basal or squamous cell carcinoma of the skin or pre-cancerous skin lesions.

   22. Has a history of cancer within the last 10 years except for basal cell or squamous cell carcinomas of the skin or in situ carcinoma of the cervix treated and considered cured.

   23. Has a history of drug abuse (defined as any illicit drug use), or a history of alcohol abuse within 2 years prior to the Screening visit.

   24. Has a severe psychiatric or neurological disorder. 25. If female, the participant is pregnant or lactating or intends to become pregnant before, during, or within 18 weeks after the last treatment visit; or intends to donate ova during such time periods.

   26. If male, the participant intends to donate sperm during or within 18 weeks after the last treatment visit.

   27. Has plans to donate germ cells, organs or bone marrow during the course of the study and within 6 months after the last injection of investigational medicinal product (IMP).

   28. Elective surgical procedure, including bone or joint surgery/ synovectomy (including joint fusion or replacement) within 12 weeks prior to baseline visit, or if the participant plans to have elective surgical procedure during the study, or within 18 weeks after the last treatment visit.

   29. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee involved in conduct of this study (eg, spouse, parent, child, sibling), or may consent under duress.

   30. Is suspected to be unable or unwilling to adequately comply with study procedures eg, language problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (31):
- Bulgaria (3):
  - Plovdiv
  - Rousse
  - Sofia
- Czechia (4):
  - České Budějovice
  - Prague
  - Uherské Hradiště
  - Zlín
- Japan (13):
  - Fukuoka, Fukuoka
  - Iizuka-shi, Fukuoka
  - Kitakyusyu-shi, Fukuoka
  - Sapporo, Hokkaido
  - Takarazuka-shi, Hyōgo
  - Morioka, Iwate
  - Kawasaki-shi, Kanagawa
  - Kumamoto, Kumamoto
  - Miyagi-gun, Miyagi
  - Nagasaki, Nagasaki
  - Sasebo-shi, Nagasaki
  - Hamamatsu, Shizuoka
  - Nishimuro-gun, Wakayama
- Poland (2):
  - Bydgoszcz
  - Torun
- Russia (4):
  - Kazan'
  - Saint Petersburg
  - Ulyanovsk
  - Voronezh
- Seoul, Gyeonggi-do, South Korea
- Spain (2):
  - A Coruña
  - Seville
- United Kingdom (2):
  - Romford, Essex
  - London, Greater London

REFERENCES:
- [Derived] Taylor PC, Saurigny D, Vencovsky J, Takeuchi T, Nakamura T, Matsievskaia G, Hunt B, Wagner T, Souberbielle B; NEXUS Study Group. Efficacy and safety of namilumab, a human monoclonal antibody against granulocyte-macrophage colony-stimulating factor (GM-CSF) ligand in patients with rheumatoid arthritis (RA) with either an inadequate response to background methotrexate therapy or an inadequate response or intolerance to an anti-TNF (tumour necrosis factor) biologic therapy: a randomized, controlled trial. Arthritis Res Ther. 2019 Apr 18;21(1):101. doi: 10.1186/s13075-019-1879-x. PMID 30999929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 28 investigative sites in Bulgaria, Czech Republic, Japan, Poland, Russian Federation, Spain and the United Kingdom from 17 December 2014 to 05 December 2016.
Pre-assignment Details: Participants with a diagnosis of moderate to severe Rheumatoid Arthritis were enrolled equally in one of 4 treatment groups: placebo or 20, 80, 150 mg/mL namilumab.
Period: Overall Study
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Started | 27 | 28 | 25 | 28
Full Analysis Set | 26 (One participant was excluded because of data collection issues.) | 28 | 24 (One participant was excluded because of data collection issues.) | 28
Completed | 15 | 18 | 18 | 14
Not Completed | 12 | 10 | 7 | 14
Not completed — Pretreatment Event/Adverse Event | 0 | 2 | 0 | 1
Not completed — Principal Investigator Discretion | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Voluntary Withdrawal | 2 | 5 | 2 | 4
Not completed — Study Termination | 7 | 2 | 5 | 8
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set includes all participants who received at least 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL | Total
Number analyzed (Participants) | 27 | 28 | 25 | 28 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.45) | 46.1 (10.07) | 49.0 (9.60) | 51.3 (14.13) | 48.4 (12.02)
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 9 | 11 | 7 | 7 | 34
  45 to 64 years | 15 | 16 | 17 | 19 | 67
  65 to 74 years | 1 | 1 | 1 | 2 | 5
  >= 75 years | 2 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 17 | 22 | 84
  Male | 4 | 6 | 8 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 0 | 4
  Not Hispanic or Latino | 22 | 22 | 21 | 23 | 88
  Unknown or Not Reported | 4 | 4 | 3 | 5 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 4 | 3 | 5 | 18
  White | 21 | 24 | 22 | 22 | 89
  Multiracial | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 2 | 1 | 1 | 1 | 5
  Czech Republic | 7 | 9 | 9 | 10 | 35
  Japan | 4 | 4 | 3 | 5 | 16
  Poland | 1 | 6 | 4 | 2 | 13
  Russia | 7 | 4 | 6 | 9 | 26
  Spain | 1 | 2 | 1 | 0 | 4
  United Kingdom | 5 | 2 | 1 | 1 | 9
Height [Mean (Standard Deviation); unit: cm] | 164.3 (10.51) | 167.7 (6.65) | 167.4 (8.36) | 166.5 (9.24) | 166.5 (8.78)
Weight [Mean (Standard Deviation); unit: kg] | 63.89 (14.511) | 70.28 (15.911) | 76.56 (18.660) | 72.23 (19.168) | 70.64 (17.499)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.75 (5.542) | 24.91 (5.210) | 27.16 (5.605) | 25.92 (6.313) | 25.41 (5.741)
BMI Categories [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 24 | 23 | 16 | 22 | 85
  >= 30 kg/m^2 | 3 | 5 | 9 | 6 | 23
Smoking classification [Count of Participants; unit: Participants]
  Participant has never smoked | 16 | 19 | 18 | 18 | 71
  Participant is a current smoker | 6 | 5 | 5 | 6 | 22
  Participant is an ex-smoker | 5 | 4 | 2 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28 C-Reactive Protein (DAS28-CRP) at Week 12
Description: The DAS28-CRP score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], general health: patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and acute phase response: C-Reactive Protein (CRP) for a total possible score of 0 (best) to approximately 10 (worst). Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicates improvement. A mixed model repeated measures (MMRM) model with main effects for study site, treatment, visit, and previously failed medication with interactions between visit and treatment, visit and previously failed medication, and visit and baseline value as a covariate and participant as a random effect with an unstructured covariance structure was used for analysis.
Time Frame: Baseline and Week 12
Population: Participants from the Full Analysis Set (FAS), all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in double-blind period up to Week 12, with data available at Baseline and Week 12 for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 24 | 25 | 22 | 26
score on a scale | -0.77 (0.294) | -1.38 (0.288) | -1.36 (0.302) | -1.69 (0.286)
Statistical Analysis 1: Comparison: Placebo vs Namilumab 20 mg/mL; Test type: Superiority or Other; p = 0.086, ANOVA — MMRM model with main effects for study site, treatment, visit, and previously failed medication with interactions between visit and treatment, visit and previously failed medication, and visit and baseline value; Baseline values were used as a covariate and participant as a random effect with an unstructured covariance structure; Least Squares (LS) Mean Difference = -0.61, 95% CI 2-sided [-1.31 to 0.09], Standard Error of Mean 0.351 — Namilumab - Placebo
Statistical Analysis 2: Comparison: Placebo vs Namilumab 80 mg/mL; Test type: Superiority or Other; p = 0.107, ANOVA — [p-value comment as in outcome 1, analysis 1]; Baseline values were used as a covariate and subject as a random effect with an unstructured covariance structure; LS Mean = -0.60, 95% CI 2-sided [-1.32 to 0.13], Standard Error of Mean 0.366 — Namilumab - Placebo
Statistical Analysis 3: Comparison: Placebo vs Namilumab 150 mg/mL; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 1, analysis 1]; Baseline values were used as a covariate and subject as a random effect with an unstructured covariance structure; LS Mean Difference = -0.92, 95% CI 2-sided [-1.61 to -0.23], Standard Error of Mean 0.347 — Namilumab - Placebo

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20), 50% (ACR 50) and 70% (ACR70) Response at Weeks 12 and 24
Description: ACR20/50/70 response is defined as a ≥20/50/70% reduction from Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), and the following:
  * Patient's Assessment of Pain over the previous 24 hours using a Visual Analog Scale (VAS); left end of the line 0=no pain to right end of the line 100=unbearable pain
  * Patient's Global Assessment of Disease Activity
  * Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity
  * Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do
  * Acute-phase reactant: C-reactive Protein (CRP).
Time Frame: Baseline and Weeks 12 and 24
Population: FAS includes all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in the double-blind period up to Week 12. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 26 | 28 | 24 | 28
percentage of participants
  ACR 20, Week 12: number analyzed (Participants) | 24 | 25 | 23 | 26
  ACR 20, Week 12 | 37.5 | 72.0 | 52.2 | 53.8
  ACR 50, Week 12: number analyzed (Participants) | 24 | 25 | 23 | 26
  ACR 50, Week 12 | 16.7 | 20.0 | 30.4 | 38.5
  ACR 70, Week 12: number analyzed (Participants) | 24 | 25 | 23 | 26
  ACR 70, Week 12 | 8.3 | 4.0 | 21.7 | 15.4
  ACR 20, Week 24: number analyzed (Participants) | 21 | 23 | 23 | 25
  ACR 20, Week 24 | 33.3 | 65.2 | 47.8 | 56.0
  ACR 50, Week 24: number analyzed (Participants) | 21 | 23 | 23 | 25
  ACR 50, Week 24 | 23.8 | 34.8 | 47.8 | 36.0
  ACR 70, Week 24: number analyzed (Participants) | 21 | 23 | 23 | 25
  ACR 70, Week 24 | 19.0 | 13.0 | 30.4 | 20.0

3. Secondary Outcome: ACR Numeric (N) Index (ACRn) at Week 12
Description: ACRn is defined as the lowest % improvement for TJC68, SJC66 and the median of 5 ACR components. These are • Patient's Assessment of Pain over previous 24 hours using a VAS; left end of line 0=no pain to right end of line 100=unbearable pain • Patient's Global Assessment of Disease Activity • Physician's Global Assessment of Disease Activity over previous 24 hours using a VAS where left end of line 0=no disease activity to right end of line 100=maximum disease activity • Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do • Acute-phase reactant: CRP. A positive % change indicates improvement. MMRM model with main effects for study site, treatment, visit, and previously failed medication with interactions between visit and treatment and visit and previously failed medication and participant used as a random effect with an unstructured covariance structure.
Time Frame: Baseline and Week 12
Population: Participants from the FAS, all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in the double-blind period up to Week 12, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 24 | 25 | 23 | 26
percentage change | -17.25 (16.469) | 3.97 (16.372) | 19.68 (16.875) | 17.14 (16.098)

4. Secondary Outcome: ACR Numeric (N) Index (ACRn) at Week 24
Description: as for outcome 3
Time Frame: Baseline and Week 24
Population: Participants from the FAS, all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in the double-blind period up to Week 12, with data available for analysis. Post-escape data is included.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 26 | 28 | 24 | 28
percentage change | 34.04 (40.248) | 35.35 (50.191) | 44.66 (38.203) | 36.57 (38.709)

5. Secondary Outcome: Change From Baseline in DAS28-CRP at Weeks 2, 6, and 10
Description: The DAS28-CRP score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], general health: patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and acute phase response: C-Reactive Protein (CRP) for a total possible score of 0 (best) to approximately 10 (worst). Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicates improvement. A MMRM model with main effects for study site, treatment, visit, and previously failed medication with interactions between visit and treatment, visit and previously failed medication, and visit and baseline value as a covariate and participant as a random effect with an unstructured covariance structure was used for analysis.
Time Frame: Baseline and Weeks 2, 6 and 10
Population: FAS includes all participants in the safety analysis set who had at least 1 valid postbaseline assessment of DAS28-CRP in the double-blind period up to Week 12. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 26 | 28 | 24 | 28
score on a scale
  Change at Week 2: number analyzed (Participants) | 26 | 28 | 23 | 28
  Change at Week 2 | -0.33 (0.236) | -0.58 (0.222) | -0.84 (0.245) | -0.95 (0.224)
  Change at Week 6: number analyzed (Participants) | 25 | 26 | 23 | 27
  Change at Week 6 | -0.70 (0.268) | -1.13 (0.256) | -1.37 (0.275) | -1.42 (0.257)
  Change at Week 10: number analyzed (Participants) | 25 | 25 | 22 | 27
  Change at Week 10 | -0.75 (0.280) | -1.19 (0.273) | -1.39 (0.289) | -1.51 (0.269)

6. Secondary Outcome: Change From Baseline in DAS28-CRP at Week 24
Description: The DAS28-CRP score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], general health: patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and acute phase response: C-Reactive Protein (CRP) for a total possible score of 0 (best) to approximately 10 (worst). Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Participants from the FAS, all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in the double-blind period up to Week 12, with data available for analysis at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 12 | 18 | 16 | 17
score on a scale | -1.75 (1.401) | -2.37 (1.083) | -2.20 (1.219) | -2.26 (0.962)

7. Secondary Outcome: Percentage of Participants With a Reduction of Pain as Measured Using a Visual Analog Scale (VAS) at Weeks 2, 12 and 24
Description: Reduction of Pain, defined as a ≥40% change from Baseline as measured using a 100 mm Visual Analog Scale (VAS); left end of the line 0=no pain to right end of the line 100=unbearable pain at weeks 2, 12 and 24.
Time Frame: Baseline and Week 2, 12 and 24
Population: Participants from the FAS, all participants in the safety analysis set who had at least 1 valid post-baseline assessment of DAS28-CRP in the double-blind period up to Week 12, with data available for analysis. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL
Number analyzed (Participants) | 26 | 28 | 24 | 28
percentage of participants
  Week 2: number analyzed (Participants) | 26 | 28 | 23 | 28
  Week 2 | 7.7 | 14.3 | 8.7 | 3.6
  Week 12: number analyzed (Participants) | 24 | 25 | 23 | 26
  Week 12 | 20.8 | 44.0 | 39.1 | 30.8
  Week 24: number analyzed (Participants) | 22 | 23 | 23 | 25
  Week 24 | 22.7 | 43.5 | 47.8 | 24.0

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug (Up to 46.4 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Placebo: Namilumab placebo-matching, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
- Namilumab 20 mg/mL: Namilumab 20 mg/mL, subcutaneous (SC) injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
- Namilumab 80 mg/mL: Namilumab 80 mg/mL, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
- Namilumab 150 mg/mL: Namilumab 150 mg/mL, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
- Placebo to Namilumab 150 mg/mL: Namilumab placebo-matching, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 12; followed by Namilumab 150 mg/mL, SC injection, every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
- Namilumab to Namilumab 150 mg/mL: Namilumab 20 or 80 mg/mL, SC injection, once on Days 1, 15, 43, 71 and every 4 weeks up to Week 12; followed by namilumab 150 mg/mL, SC injection, every 4 weeks up to Week 24. All participants were on a stable dose of methotrexate tablets (15-25 mg weekly) and folic acid (at least 5 mg/week) orally throughout the duration of the study.
Arm/Group | Placebo | Namilumab 20 mg/mL | Namilumab 80 mg/mL | Namilumab 150 mg/mL | Placebo to Namilumab 150 mg/mL | Namilumab to Namilumab 150 mg/mL
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 1/25 | 1/28 | 0/12 | 4/24
Other Adverse Events (participants affected / at risk) | 9/27 | 13/28 | 12/25 | 12/28 | 5/12 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Namilumab 20 mg/mL (N=28) | Namilumab 80 mg/mL (N=25) | Namilumab 150 mg/mL (N=28) | Placebo to Namilumab 150 mg/mL (N=12) | Namilumab to Namilumab 150 mg/mL (N=24)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Namilumab 20 mg/mL (N=28) | Namilumab 80 mg/mL (N=25) | Namilumab 150 mg/mL (N=28) | Placebo to Namilumab 150 mg/mL (N=12) | Namilumab to Namilumab 150 mg/mL (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 7 | 2 | 5 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.